CLINICAL TRIAL: NCT04317651
Title: Crizotinib in ALK Rearranged Non-small-cell Lung Cancer
Acronym: SPECIALK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Other Study IDs: SPECIALK
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer; Advanced Cancer; Metastatic Cancer
Keywords: crizotinib; Non Small Cell Lung Cancer; Metastatic Cancer; Advanced Cancer; NSCLC; ALK positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, observational, retrospective cohort study aimed at assessing the efficacy and safety of crizotinib in ALK positive NSCLC treated in real life setting.

DETAILED DESCRIPTION:
Primary efficacy objective:

To assess the efficacy of crizotinib in real life setting

Secondary objectives:

1. To evaluate the therapeutic response to crizotinib-based treatment
2. To identify additional biomarkers selectively present in the ALK positive population
3. To assess the safety of crizotinib (250 mg/bid) in the treatment of NSCLC in real life setting

Non-small-cell Lung Cancer (NSCLC) remains the leading cause of cancer death in Western Countries. Identification of anaplastic lymphoma kinase (ALK) gene rearrangements reinforced the role of targeted therapies in lung cancer. The EML4-ALK fusion gene is detected in 3-7% of patients with adenocarcinomas of the lung and is associated with specific clinical pathological features, including young age, absent or minimal smoking history and adenocarcinoma histology. However, such clinical features do not properly select patients for ALK inhibitors (ALK-Is) and, consequently, molecular testing is mandatory. Indeed, current guidelines recommend to test ALK rearrangements at diagnosis all patients with advanced lung adenocarcinoma, due to immediate therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and Females aged 18 years with diagnosis of advanced or metastatic NSCLC
* 2. Former participation in the Italian NPU program between December 2010 - April 2013 or receiving crizotinib according to 648 legislative Decrete from April 2013 to February 2015 and thereafter in clinical practice up to December 31st, 2017.
* 3. Ascertained compliance to the Crizotinib therapy as prescribed by the relevant physician
* 4. ALK rearrangement report including details of method and cutoff used for ALK testing
* 5. Data on prior therapies
* 6. Data on toxicity
* 7. Data on crizotinib therapy efficacy including response to the therapy and survival
* 8. Data on site of metastases
* 9. Availability of archival tissue (not mandatory)
* 10. Signed Informed Consent for alive and contactable patients

Exclusion Criteria:

* 1. Lack of clinical data
* 2. No evidence of ALK rearrangemement
* 3. Early death defined as fatal outcome within 30 days since the first crizotinib dose
* 4. Absence of any radiological assessment
* 5. No data on crizotinib efficacy including survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with crizotinib at the standard doses of 250 mg/bid. Based on the total number of patients treated with Crizotinib in the NPU program (approximately 900) as well as on the clinical experience, the investigators expect that almost 500 patients will enter this study and that tumor biopsies will be available on approximately 100 patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Sistematic review of medical records | Six months
  To assess the overall efficacy of crizotinib (250 mg/bid) in terms of Response rate, Progression-Free Survival and Overall Survival in the treatment of NSCLC in real life setting. Median PFS, as reported by a recent metanalysis, is 9.4 months (first and second line together) corresponding to a 12 months PFS rate of about 40%. The analysis of 500 patients will allow to estimate the median PFS with a semi-width 95% confidence interval of 1.2 months. OS will be calculated from the first day of treatment until the date of death from any cause. Any patient not known to have died at the time of data analysis will be censored at the time of the last recorded date on which the patient was known to be alive. Time to events will be summarized using Kaplan-Meier estimation.
  ORR, defined as the proportion of patients with a best overall response of either Complete response or Partial response, will be calculated based on disease status evaluated by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Secondary Objectives | Six months
  1. To define clinical and biological characteristics of patients not responding to crizotinib therapy at the first tumor assessment versus individuals with complete or deep partial response (> 50% reduction in the sum of target lesions)
  2. To define additional biomarkers selectively present in the ALK positive population
  3. To explore outcome of individuals with brain metastases
  4. To define timing of local ablative therapy in presence of brain metastas

CONTACTS AND LOCATIONS:
Locations (23):
- Italy (23):
  - Ospedale Versilia, Camaiore, Lucca
  - A.O. San Gerardo, Monza, Milano
  - Ospedale Oncologico Regionale - Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, Potenza
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, Ravenna
  - A.O.U. San Luigi Gonzaga, Orbassano, Torino
  - Sacro Cuore- Don Calabria Hospital, Negrar, Verona
  - Azienda Ospedaliera di Rilievo Nazionale "S.G. Moscati", Avellino
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AO Papardo, Messina
  - Istituto Europeo di Oncologia, Milan
  - A.O.R.N dei Colli - Ospedale Monaldi, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Ospedale Giovanni Paolo II ASL-2 Olbia, Olbia
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera-Universitaria di Parma, Parma
  - Ospedale Santa Maria della Misericordia - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale di Ravenna, Ravenna
  - IRCCS- Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Universitario "Campus Biomedico" di Roma, Roma
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - ASST Sette Laghi "Ospedale di Circolo e Fondazione Macchi", Varese
  - Policlinico 'G.B.Rossi' Borgo Roma - Azienda Ospedaliera Universitaria Integrata (Giampaolo Tortora), Verona

IPD SHARING:
Plan to Share IPD: Undecided